CLINICAL TRIAL: NCT01296295
Title: Effectiveness of Regular Reporting of Spirometric Results Combined With a Smoking Cessation Advice by a Primary Care Physician on Smoking Quit Rate in Adult Smokers: a Randomized Controlled Trial.
Brief Title: Effectiveness of Regular Reporting of Spirometric Results on Smoking Quit Rate.
Acronym: ESPIROTAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Catalan Institute of Health (Other Government); Research Support Unit Metropolitana Nord, Barcelona, Spain (Unknown)
Responsible Party: Maria del Mar Rodriguez Alvarez, Catalan Health Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P10/40.; Jordi Gol i Gurina Foundation (Registry Identifier: P10/40)
Record Dates: First submitted 2010-07-30; First posted 2011-02-15 (Estimated); Last update posted 2011-02-15 (Estimated); Status verified 2011-02

CONDITIONS: Smoking Cessation; COPD
Keywords: smoking cessation advice; spirometry; primary health care
MeSH Terms: conditions — Smoking Cessation; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Spirometry and lifestyle counseling (Experimental): Intervention group: The intervention is to give brief structured smoking cessation advice combined with a detailed and structured discussion of the spirometric results.
  Interventions: Behavioral: Lifestyle counseling and spirometry
- Lifestyle counseling (No Intervention): No intervention group: the patients of the control group will receive a brief structured smoking cessation advice.
  Interventions: Behavioral: Smoking cessation advice

INTERVENTIONS:
Behavioral: Lifestyle counseling and spirometry — The patients of the intervention group will be given a brief structured smoking cessation advice by their primary care physician combined with a detailed and structured discussion of the spirometry results.
  Arms: Spirometry and lifestyle counseling
Behavioral: Smoking cessation advice — Brief smoking cessation advice
  Arms: Lifestyle counseling

SUMMARY:
The purpose of this study is to evaluate the effectiveness of regular reporting of spirometric results combined with smoking cessation advice on smoking quit rate in adult smokers in primary care.

Hypothesis: In adult smokers, regular reporting of spirometric test results in addition with smoking cessation advice will increase smoking quit rate.

Expected outcome: increase of smoking cessation rate .

DETAILED DESCRIPTION:
Design: Intervention study with two randomized arms in 5 primary care centers of two health areas.

Study population: 466 smokers over the age of 18 consulting their primary care physician for any reason and who do not fulfil the exclusion criteria.

Measurements and interventions: The study data will be collected using a structured questionnaire and data collection sheets specifically designed for the study The structured questionnaire will include the following data: sociodemographics, clinical history, smoking habit, respiratory symptomatology, smoking dependence test and smoking cessation motivation test.

The data collection sheets will include information related to the spirometric results, peak expiratory flow rate and the carbon monoxide test when performed.

On visit 0, the primary care physician will give a brief structured smoking cessation advice to all patients combined with a detailed and structured discussion of the spirometric results. After this visit the patients will be randomised in two arms (control and intervention groups).

Randomisation will be performed using a computer programme.

Randomisation will be carried out by the Coordinating Centre.

Both groups will be followed up by telephone at three (visit 1) and six months (visit 2) and at one-year (visit 3) and two-year(visit 4).

During the follow up visits brief structured smoking cessation advice will be reinforced in the control group but the spirometric results will not be discussed. In the intervention group brief structured smoking cessation advice will be reinforced with a detailed structured reminder discussion of the results obtained from the spyrometry of visit 0.

Follow up visits 1 and 2 will be undertaken by telephone and the patients will be asked about their smoking habit and will be given a brief questionnaire.

One month before visits 3 and 4 both groups will undergo the same series of tests performed prior to visit 0 with the exception of the peak expiratory flow rate. Spirometry will be done only in the intervention group.

On visits 3 and 4, the same intervention will be done. On both visits 3 and 4 all the participants who report smoking withdrawal will undergo the carbon monoxide test.

ELIGIBILITY:
Inclusion Criteria:

* All adult smoker population over the age of 18 years attended by their primary care physician for any reason and who do not fulfil exclusion criteria

Exclusion Criteria:

* Previous diagnosis of COPD by spirometry.
* Patients contraindicated to undertake spirometry.
* Patients without a telephone.
* Patients with communication difficulties: cognitive and/or sensorial deterioration, language.
* Patients with severe disease of poor prognosis (life expectancy of less than one year).
* Patients with another respiratory disease: asthma, COPD, neoplasm of the respiratory tract, pulmonary thromboembolism, pulmonary tuberculosis, interstitial diseases.
* Patients who do not give written informed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 466 (Actual)
Dates: Start 2005-01; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Smoking abstinence: self reported abstinence (12 or more months smoking free. | 24 months after last recruitment
  Smoking cessation confirmed by air carbon monoxide concentration. Safety Issue?: (FDAAA) No

CONTACTS AND LOCATIONS:
Overall Officials: Mar Rodriguez, Principal Investigator — Institut Catalá de la Salut
Locations (1):
- Jordi Gol i Gurina Foundation, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Rodriguez-Alvarez M, Toran-Monserrat P, Munoz-Ortiz L, Negrete-Palma A, Montero-Alia JJ, Jimenez-Gonzalez M, Zurilla-Leonarte E, Marina-Ortega V, Olle-Borque M, Valentin-Moya E, Cortada-Cabrera A, Tena-Domingo A, Martinez-Gonzalez S, Vila-Palau V, Ramos-Ordonez A, Rotllant-Estelrich G, Forcada-Vega C, Borrell-Thio E. Effectiveness of regular reporting of spirometric results combined with a smoking cessation advice by a primary care physician on smoking quit rate in adult smokers: a randomized controlled trial. ESPIROTAB study. BMC Fam Pract. 2011 Jun 28;12:61. doi: 10.1186/1471-2296-12-61. PMID 21708047